CLINICAL TRIAL: NCT06339476
Title: Exploring the Complex Links Between Menstrual Irregularity and Cellular Markers: A Focus on the Apoptosis Marker M30, the Endothelial Function Marker Asymmetric Dimethylarginine and Malondialdehyde
Brief Title: Exploring the Complex Links Between Menstrual Irregularity and Cellular Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Dilara Ulger Ozbek, Ph.D, lecturer, Cumhuriyet University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Dilara ÜLGER ÖZBEK
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Menstrual Irregularity; Menstrual Cycle Abnormal
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Intervention Model Description: In the overall study population of 56 subjects recruited from, Sivas Cumhuriyet University Faculty of Medicine Research and Practice Hospital, Gynecology and Obstetrics Clinic, divided into two groups: irregular menstrual cycle (n=28) and regular menstrual cycle control group (n=28). While those who met the criteria for menstrual irregularity were included, those with another gynecological disease (PCOS, endometriosis, etc.) and additional diseases (diabetes, insulin resistance, cancer, heart disease, etc.) were excluded from the study. All participants provided written informed consent before participating in the study. Participants were asked to report the average length of their menstrual cycle over the past six months, as well as the consistency of cycle length. Menstrual regularity was assessed by self-report using a standardized questionnaire.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serum ADMA, MDA and M30 levels mesurment (Experimental): With the permission of the participants, 7 ml of venous, fasting blood samples were collected during the early follicular phase. In the blood serum of the participants, M30, ADMA, and MDA levels were measured by using commercial ELISA test kits.
  Interventions: Diagnostic Test: Serum ADMA, MDA and M30 levels mesurment
- diagnosis of the study group (No Intervention): Determination of the patient and control group to be included in the study group by the relevant gynecologist.

INTERVENTIONS:
Diagnostic Test: Serum ADMA, MDA and M30 levels mesurment — Blood samples collected from patienst, only 7 mL
  Other Names: Taking a blood samples
  Arms: Serum ADMA, MDA and M30 levels mesurment

SUMMARY:
A cross-sectional study design was employed, involving 56 premenopausal participants with ages ranging from 20 to 49 years. Serum samples were collected during the early follicular phase, and levels of some biochemicals parameters analyzed.

DETAILED DESCRIPTION:
A cross-sectional study was conducted to investigate the potential relationship between menstrual regularity and the apoptosis marker caspase-cleaved cytokeratin 18 fragment (M30), Asymmetric dimethylarginine (ADMA), and Malondialdehyde (MDA) levels. The investigators screened 80 participants who applied for menstrual irregularity between 2023 February and 2024 March and, in addition to menstrual irregularities, 24 individuals with additional gynecological conditions such as polycystic ovary syndrome (PCOS) and endometriosis were excluded from the study. In the overall study population of 56 subjects aged 20-49 were recruited from, Sivas Cumhuriyet University Faculty of Medicine Research and Practice Hospital, Gynecology and Obstetrics Clinic. Participants were divided into two groups: irregular menstrual cycle (28 participants) and regular menstrual cycle control group (28 participants). While those who met the criteria for menstrual irregularity were included, those with another gynecological disease (PCOS, endometriosis, etc.) and additional diseases (diabetes, insulin resistance, cancer, heart disease, etc.) were excluded from the study. All participants provided written informed consent before participating in the study. The study protocol was approved by the Sivas Cumhuriyet University, Clinical Research Ethics Committee Chairman, 2023-02/06. All procedures were performed in accordance with the ethical standards laid down in the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Menstrual Irregularity
* Being over 18 years of age and not distinguished by age.

Exclusion Criteria:

* Another gynecological disease (PCOS, endometriosis, etc.) and additional diseases (diabetes, insulin resistance, cancer, heart disease, etc.)

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
ADMA, M30 and MDA levels mesurment in the blood serum to compare between patient and control. | not measured in time frame. general (one day)
  ADMA, M30 and MDA levels mesured in the blood serum. The most common side effect when blood is taken from the patient is slight bruising and swelling in the arm due to needle sticking. There will be no other serious side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University Hospital, Sivas, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study will be opened to researchers after it is published internationally